CLINICAL TRIAL: NCT03847116
Title: Association of Light-to-moderate Alcohol Consumption With Risk of Type 2 Diabetes Mellitus in Individuals With Nonalcoholic Fatty Liver Disease
Brief Title: Alcohol Consumption and Type 2 Diabetes Mellitus Risk in Nonalcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LHNAFLD 2018-V1.0
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Nonalcoholic Fatty Liver Disease; Light-to-moderate Alcohol Consumption; Type2 Diabetes Mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explored the cross-sectional and prospective associations between light-to-moderate alcohol consumption (LMAC) and risk of type 2 diabetes mellitus (T2DM) in individuals with nonalcoholic fatty liver disease (NAFLD).

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or above
2. undergoing annual health examinations in 2009 in Zhenhai Lianhua Hospital, Ningbo, China.
3. informed about the study

Exclusion Criteria:

1. female participants;
2. missing data on ultrasound, alcohol consumption, and T2DM status;
3. alcohol consumption > 210 g per week, and binge drinkers;
4. with evidence of other liver diseases including viral hepatitis, autoimmune hepatitis, and drug-induced liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive Chinese adults underwent annual health examinations in 2009 were enrolled in the cohort study. Follow-up between 2009 and 2018 were obtained in Zhenhai Lianhua Hospital, Ningbo.
Sampling Method: Non-Probability Sample
Enrollment: 14014 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Light-to-moderate alcohol consumption (LMAC) and risk of prevalent type 2 diabetes mellitus (T2DM) | cross-sectional analyses in 2009
  Fatty liver was assessed by ultrasound. T2DM was defined as the presence of any of the following conditions based on American Diabetes Association criteria: (1) fasting plasma glucose (FPG) ≥ 7.0 mmol/L; (2) hemoglobin A1c (HbA1c) ≥ 6.5%; (3) self-reported clinician-diagnosed T2DM.

SECONDARY OUTCOMES:
LMAC and incident risk of T2DM | 9-year cohort observation
  Fatty liver was assessed by ultrasound. T2DM was defined as the presence of any of the following conditions based on American Diabetes Association criteria: (1) fasting plasma glucose (FPG) ≥ 7.0 mmol/L; (2) hemoglobin A1c (HbA1c) ≥ 6.5%; (3) self-reported clinician-diagnosed T2DM.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Xu L, Xie J, Chen S, Chen Y, Yang H, Miao M, Zhu Z, Li Y, Yu C, Xu C. Light-to-Moderate Alcohol Consumption Is Associated With Increased Risk of Type 2 Diabetes in Individuals With Nonalcoholic Fatty Liver Disease: A Nine-Year Cohort Study. Am J Gastroenterol. 2020 Jun;115(6):876-884. doi: 10.14309/ajg.0000000000000607. PMID 32282335